CLINICAL TRIAL: NCT01191385
Title: Non Interventional Study in Patients With Diagnosis of HCC in Whom a Decision to Treat With Sorafenib Has Not Been Made at Time of Study Enrollment
Brief Title: GIDEON Non-Nexavar Arm - HCC Patients Who Are Treated With Any Therapy Other Than Nexavar at Individual Study Start
Status: Withdrawn | Type: Observational
Why Stopped: Study is officially cancelled bevore FPFV.
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 14611; NX0901
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2015-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; Liver cancer; Cancer of liver; Cancer, liver; Hepatic cancer; Cancer, hepatic; Carcinoma, hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Any treatment for unresectable HCC as chosen by the physician

INTERVENTIONS:
Drug: Any treatment for unresectable HCC as chosen by the physician — Only those patient are allowed to be enrolled that receive any HCC treatment for unresectable HCC as chosen by the physician except sorafenib. During the course of the study, each treatment is allowed.

SUMMARY:
This study is an international prospective, open-label, multi-center, non-interventional study. The protocol will allow enrollment of all patients with diagnosis of HCC in whom a decision to treat with sorafenib has not been made at time of study enrollment. All patients will be followed-up until withdrawal of consent, lost to follow-up, death, or the end of the study. Detailed information concerning the past medical/surgical history, performance status, methods of diagnosis and staging, etc. of patients with HCC will be collected, and practice patterns of the physicians involved in the care of patients with HCC under real-life conditions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with histologically/cytologically documented or radiographically diagnosed HCC in whom a decision to treat with sorafenib has not been made at this time. Radiographic diagnosis needs typical findings of HCC by radiographic method i.e. on multi-dimensional dynamic CT, CT hepatic arteriography (CTHA)/CT arterial portography (CTAP) or MRI.
* Patients must have signed an informed consent form
* Patients must have a life expectancy of at least 8 weeks

Exclusion Criteria:

* Patients in whom a decision to treat with sorafenib is made at time of study start
* Patients who have received sorafenib in the past or are currently treated with sorafenib
* Hospice patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC in whom a decision to treat with sorafenib has not been made at time of study enrollment and who were never treated with sorafenib in the past
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determination of 'real-life' practice patterns of physicians involved in the care of patients with HCC (collection of data on treatments prescribed as well as demographic data and data on the entire medical history) | up to 3,3 years
Evaluation of patient demographics, disease characteristics, methods of patient evaluation, diagnosis and follow-up of patients with HCC, regionally and globally (collection of data on demographics, medical history, diagnostic measurements, follow-up) | up to 3,3 years

SECONDARY OUTCOMES:
Evaluation of natural course and outcomes of patients with HCC (collection of data of disease status during the course of the study and the outcome of treatment) | up to 3,3 years
Evaluation of treatment modalities that are used for patients with HCC during the course of their disease (collection of data of all treatments prescribed during the course of the study) | up to 3,3 years
Evaluation of safety and tolerability of treatments that are used for patients with HCC (collection of all adverse events) | up to 3,3 years
Evaluation efficacy parameters including: overall survival (OS), progression-free survival (PFS), time to progression (TTP), response rate (RR) and stable disease (SD) rate of the various interventions employed in the care of patients with HCC | up to 3,3 years
To evaluate the comorbidities in patients with HCC and their influence on treatment options and outcome (collection of data on concomitant diseases) | up to 3,3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (24):
- United States (24):
  - Multiple Locations, Arkansas
  - Multiple Locations, California
  - Multiple Locations, Colorado
  - Multiple Locations, District of Columbia
  - Multiple Locations, Florida
  - Multiple Locations, Georgia
  - Multiple Locations, Illinois
  - Multiple Locations, Indiana
  - Multiple Locations, Iowa
  - Multiple Locations, Kentucky
  - Multiple Locations, Louisiana
  - Multiple Locations, Maryland
  - Multiple Locations, Massachusetts
  - Multiple Locations, Michigan
  - Multiple Locations, Minnesota
  - Multiple Locations, Missouri
  - Multiple Locations, New Hampshire
  - Multiple Locations, New Jersey
  - Multiple Locations, New York
  - Multiple Locations, Oregon
  - Multiple Locations, Pennsylvania
  - Multiple Locations, South Carolina
  - Multiple Locations, Texas
  - Multiple Locations, Virginia